CLINICAL TRIAL: NCT06869837
Title: Effects of External Oblique Intercostal Plane Block Applied in Laparoscopic Cholecystectomy Surgery on Intraoperative Opioid ConsumptionDetermined by ANI (Analgesia Nociceptive Index) and Postoperative Analgesia Quality Guide; A Randomized Controlled Trial
Brief Title: EOIPB in Laparoscopic Cholecystectomy: Impact on Opioid Consumption Guided by ANI and Analgesia Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OMUKAEK 2024/269
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-04

CONDITIONS: Pain Management; Laparoscopic Cholecystectomy Surgery
Keywords: external oblique intercostal plane block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EOİPB (Active Comparator): Bilateral External oblique intercostal plane block will be applied 45 minutes before surgery.
  Interventions: Other: Group EOİPB
- Group Control (No Intervention): No intervention will be made in this group.

INTERVENTIONS:
Other: Group EOİPB — Bilateral external oblique intercostal plane block under USG guidance will be applied 45 minutes before cholecystectomy surgery.
  Arms: Group EOİPB

SUMMARY:
The aim of the study was to evaluate the response of regional anesthesia to remifentanyl consumption in patients undergoing laparoscopic cholecystectomy surgery.

DETAILED DESCRIPTION:
Routine anesthesia and analgesia protocol will be applied to all participants. The study aims to evaluate the remifentanyl consumption of the participants by dividing them into two groups as those with and without block and then performing their monitoring (pulse, mean arterial pressure with noninvasive measurement, oxygen saturation, Analgesia Nociception Index, Bispectral index). Remifentanil level will be adjusted according to the ANI value. The target is to keep the ANI between 50-70.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will undergo elective laparoscopic cholecystectomy surgery,
* Age 18-70,
* ASA I-II physical status,
* Body mass index (BMI) < 35 kg/m²,
* Participants who have written consent to participate in the study

Exclusion Criteria:

* Participants with routine analgesic consumption,
* Those with coagulopathy,
* Those with a history of local anesthetic allergy,
* Those with cardiac arrhythmia and pacemaker,
* ASA III and above, Those with dementia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Intraoperative opioid consumption | During surgery
  Total amount of remifentanil consumed during cholecystectomy surgery

SECONDARY OUTCOMES:
Numeric rating scale for postoperative pain intensity | up to 24 hours (Will be evaluated at 1, 3, 6, 9, 12, 18, 24 hours)
  Evaluated with a Numerical rating scale (NRS) from 0 to 10. (0=no pain; 10=worst imaginable pain)
Quality of Recovery - 15 score | Postoperative 24th hour
  The impact of surgical and anesthetic interventions on perioperative quality of life and ability to resume routine life activities will be assessed using the Quality of Recovery (QoR) tool. Each question is scored between 0 and 10. The survey result varies between 0-150 points based on the answers given by the patients. Higher scores indicate better recovery.
Fentanyl consumption at 30 minutes after arrival in the PACU(post anesthesia care unit) | 30 minutes
  Evaluated with a NRS from 0 to 10 and fentanyl will be administered when NRS is 4 and above. Fentanyl consumed will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: HALE K CELIK, Study Director — SAMSUN UNİVERSITY
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, İ̇lkadim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/ or analysed during the current study are available from the corresponding author on reasonable request.